CLINICAL TRIAL: NCT00375687
Title: Investigation of Early Hormonotherapy Efficacy of High Risk Patients for Progression of Prostate Cancer After Radical Prostatectomy
Brief Title: Investigation of Early Hormonotherapy Efficacy of Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaunas University of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMU-Urol1
Record Dates: First submitted 2006-09-12; First posted 2006-09-13 (Estimated); Last update posted 2006-09-13 (Estimated); Status verified 2005-11

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Triptorelin Pamoate

INTERVENTIONS:
Drug: Triptorelin

SUMMARY:
The purpose of this study is to determine whether early hormonotherapy is effective in the treatment of high risk prostate cancer patients after radical prostatectomy.

DETAILED DESCRIPTION:
The primary purpose of this study is to evaluate the hypothesis, that early administration of adjuvant hormonotherapy (triptorelin) can prolong survival data for high risk patients. Control group (randomised study) will be treated with hormonotherapy, when PSA recidive appear (on demand treatment). Secondary purposes will be to compare PSA dinamics and quality of life data in the groups.

ELIGIBILITY:
Inclusion Criteria:

* preoperative PSA>20ng/ml
* postoperative PSA >0.2 ng/ml
* Gleason > 7
* pT3b
* signated infomed consent

Exclusion Criteria:

* neoadjuvant hormonaltherapy before RP
* R1 RP
* N+ RP
* unstable cncomitant conditions

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61
Dates: Start 2005-08; Study Completion 2020-01

PRIMARY OUTCOMES:
Survival

SECONDARY OUTCOMES:
PSA dinamics
quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Mindaugas Jievaltas, MD, PhD, Principal Investigator — Urology dep. of Kaunas University of Medicine
Locations (1):
- Urology dep. of Kaunas University of Medicine, Kaunas, Lithuania